CLINICAL TRIAL: NCT06972173
Title: By the WHO and ICMJE for Studies With a Study Start Date That is Before June 1, 2024
Brief Title: SHORT-TERM EFFECTS OF DEEP BREATHING AND PROGRESSIVE MUSCLE RELAXATION EXERCISES ON MUSCULOSKELETAL PAIN AND WELL-BEING IN HIGH SCHOOL STUDENTS
Acronym: Deep breathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Burcu Özüberk, Principal Investigator, PT, PhD, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202300022
Record Dates: First submitted 2025-04-29; First posted 2025-05-14 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: Deep Breathing Maneuver; PROGRESSIVE MUSCLE RELAXATION EXERCISES
Keywords: Deep breathing exercises; progressive muscle relaxation exercises; high school students; musculoskeletal pain; well-being
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Exercise and control groups/RCT
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXERCISE GROUP (Experimental): The exercise program consisting of deep breathing and progressive muscle relaxation exercises was applied to the students in the exercise group. The first exercise session was started the day after the training about the study. During the study period, the program was started at the end of school hours of high school students for a total of 20 sessions (4 weeks, every weekday), each session lasting 30 minutes. The sessions started with deep breathing exercises, continued with progressive muscle relaxation exercises, and ended with deep breathing exercises.
  For deep breathing exercises, students were asked to place their dominant hand on their abdomen and non-dominant hand on their chest in the semi-fowler position. Afterwards, they were instructed to breath deeply through their nose for 4 seconds and exhale through their mouth for 8 seconds. These exercises were performed as 4 repetitions with 2 minutes rest time between the exercises. When the deep breathing exercise
  Interventions: Other: DEEP BREATHING AND PROGRESSIVE MUSCLE RELAXATION EXERCISES
- CONTROL GROUP (No Intervention): no treatment was applied to student in the control group.

INTERVENTIONS:
Other: DEEP BREATHING AND PROGRESSIVE MUSCLE RELAXATION EXERCISES — For deep breathing exercises, students were asked to place their dominant hand on their abdomen and non-dominant hand on their chest in the semi-fowler position. Afterwards, they were instructed to breath deeply through their nose for 4 seconds and exhale through their mouth for 8 seconds. These exercises were performed as 4 repetitions with 2 minutes rest time between the exercises. When the deep breathing exercises were finished, the students lay on their backs and rested for 1 minute and then progressive muscle relaxation exercise was started (10,11).
  For the progressive muscle relaxation exercise, the students were asked to contract and then relax the right foot, left foot, right leg, left leg, hip, abdominal muscles, chest muscles and back muscles, right hand, left hand, right arm, left arm, neck and shoulders, and facial muscles respectively. Respectively, from bottom to top, all the major muscles are contracted while inhaling deeply and slowly, and relaxed and r
  Arms: EXERCISE GROUP

SUMMARY:
Exam stress in high school students, long hours of studying in the static posture, and lack of physical activity habits can cause physical and psychological discomfort in them. This discomfort can be physically seen as musculoskeletal pain, while as psychologically it can be observed as a decrease in well-being. This situation can cause the acute onset of musculoskeletal pain in students to become chronic with a decrease in well-being. On the contrary, we can observe an increase in musculoskeletal pain due to stress that may occur due to a decrease in well-being.

Musculoskeletal pain is a condition that is not fatal but severely impairs health and well-being (1). According to the biopsychosocial model, pain occurs in a complex interaction between biological, psychological and social factors (2). Therefore, pain is both a subjective experience and a physical sensation with large individual differences (3). Relaxation is now a non-pharmacological intervention that has been increasingly accepted in recent years to reduce and cope with pain (4). A person who is relaxed usually has a physical and psychological well-being and feelings of calmness (5). With relaxation exercises, the person starts to reduce anxiety level by coping with stress (6). In addition to relaxation techniques, deep breathing exercise, also known as diaphragmatic breathing, is a technique based on the idea that mind and body integration provides relaxation (7). Breathing exercises are easy to learn and practice and benefit can be obtained from deep breathing exercises performed in a short time (5 minutes of practice may be sufficient) (8). In studies in which both techniques were used separately, it was reported to provide physical and psychological relaxation.

The unique aspect of this study is the investigation of the effects of both techniques on pain and well-being in high school students using both techniques simultaneously.

For this purpose, we planned to investigate the short-term effects of deep breathing and progressive muscle relaxation exercises on musculoskeletal pain and well-being in high school students.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were voluntary acceptance to participate in the exercise program with parental consent, the absence of an orthopedic, neurological or psychiatric disorder that would affect participation in exercises, and full participation in exercise sessions.

Exclusion Criteria:

* Those who did not meet the inclusion criteria and did not voluntarily agree to participate in the study

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
musculoskeletal pain | From enrollment to the end of treatment at 4 weeks
  Cornell Musculoskeletal Disorder Questionnaire (CMDQ): The scale was adapted into Turkish by Erdinç et al. in 2008. This scale assesses the frequency and severity of pain, soreness or discomfort in 11 different body parts (neck, shoulder, back, upper arm, waist, forearm, wrist, hip, upper leg, knee and lower leg) in the last 7 days and whether it interferes with work. Weight scores are calculated according to the answers given for frequency, severity and inability to work.The frequency of pain, aching or discomfort was graded from never (0) to many times every day (4); the severity was graded from mildly severe (1) to very severe (3); and the effect on work performance was graded from never interfered (1) to very much interfered (3). The weighted score for each body part takes a value between 0 and 90.

SECONDARY OUTCOMES:
WELL-BEING | From enrollment to the end of treatment at 4 weeks
  Well-being Star Scale (WSS): It is a questionnaire developed by Korkut and Owen in 2016 at the university. The first dimension 'making sense of life and being goal-oriented' consists of seven items (1, 6, 11, 16, 21, 23, 24). The second dimension 'cognitive dimension' consists of four items (2, 7, 12, 17). The third dimension, 'emotional dimension', consists of five items (3, 8, 13, 18, 22). The fourth (4, 9, 14, 19) and fifth (5, 10, 15, 20) dimensions consist of four items each and are named as 'physical dimension' and 'social dimension' respectively. The items are scored using a five-point Likert scale. The scores that can be obtained from the scale vary between 24-120 and the higher the score, the more positive the individual's well-being is interpreted.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırklareli ANATOLIA HIGH SCHOOL, Kırklareli, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: start date: 24,April, 2025 end date: 24, june, 2025